CLINICAL TRIAL: NCT01828697
Title: Low-molecular-weight Heparin to Prevent Recurrent VTE in Pregnancy: a Randomized Controlled Trial of Two Doses
Brief Title: Comparison of Low and Intermediate Dose Low-molecular-weight Heparin to Prevent Recurrent Venous Thromboembolism in Pregnancy
Acronym: Highlow
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Netherlands Organisation for Scientific Research (Other Government); Aspen Pharma (Unknown); CHU of Saint Etienne: French Ministry of Health Grant (sponsor of the French part of the study) (Unknown); Rotunda Hospital: Definitive Interventions and Feasibility Awards (DIFA) 2017 (sponsor of the Irish part of the study)) (Unknown)
Responsible Party: Principal Investigator, S. Middeldorp, prof.dr. S. Middeldorp, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Highlow study; 2012-001505-24 (EudraCT Number); NL40326.018.12 (Other: CCMO); NTR3894 (Registry Identifier: Netherlands Trial Register)
Record Dates: First submitted 2013-04-05; First posted 2013-04-11 (Estimated); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Deep Venous Thrombosis; Pulmonary Embolism
Keywords: Low-molecular-weight heparin; Pregnancy; Venous thrombosis
MeSH Terms: conditions — Venous Thrombosis; Pulmonary Embolism | interventions — Nadroparin; Enoxaparin; Dalteparin; Tinzaparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low dose LMWH (Active Comparator): Fixed low dose low-molecular-weight heparin:
  * Fixed low dose nadroparin, or;
  * Fixed low dose enoxaparin, or;
  * Fixed low dose dalteparin, or;
  * Fixed low dose tinzaparin.
  Interventions: Drug: Low dose nadroparin; Drug: Low dose enoxaparin; Drug: Low dose dalteparin; Drug: Fixed low dose tinzaparin
- Intermediate dose LMWH (Active Comparator): Intermediate dose low-molecular-weight heparin. Dosing is weight-adjusted according to the protocol.
  * Intermediate dose nadroparin, or;
  * Intermediate dose enoxaparin, or;
  * Intermediate dose dalteparin, or;
  * Intermediate dose tinzaparin.
  Interventions: Drug: Intermediate dose nadroparin; Drug: Intermediate dose enoxaparin; Drug: Intermediate dose dalteparin; Drug: Intermediate dose tinzaparin

INTERVENTIONS:
Drug: Low dose nadroparin — Fixed low dose nadroparin:
  * < 100 kg: 2850 IU subcutaneously once-daily
  * 100 kg and above: 3800 IU subcutaneously once-daily
  Other Names: nadroparin; Fraxiparin
  Arms: Low dose LMWH
Drug: Intermediate dose nadroparin — Intermediate weight-adjusted dose nadroparin:
  * < 50 kg: 3800 IU subcutaneously once-daily;
  * 50 to < 70 kg: 5700 IU subcutaneously once-daily;
  * 70 to < 100 kg: 7600 IU subcutaneously once-daily;
  * 100 kg or above: 9500 IU subcutaneously once-daily.
  Other Names: nadroparin; Fraxiparin
  Arms: Intermediate dose LMWH
Drug: Low dose enoxaparin — Fixed low dose enoxaparin:
  * < 100 kg: 40 mg subcutaneously once-daily
  * 100 kg and above: 60 mg subcutaneously once-daily
  Other Names: enoxaparin; Clexane
  Arms: Low dose LMWH
Drug: Intermediate dose enoxaparin — Intermediate weight-adjusted dose enoxaparin:
  * < 50 kg: 60 mg subcutaneously once-daily, or;
  * 50 kg to < 70 kg: 80 mg subcutaneously once-daily, or;
  * 70 kg to < 100 kg: 100 mg subcutaneously once-daily, or;
  * 100 kg or above: 120 mg subcutaneously once-daily.
  Other Names: enoxaparin; Clexane
  Arms: Intermediate dose LMWH
Drug: Low dose dalteparin — Fixed low dose dalteparin:
  * < 100 kg: 5000 IU subcutaneously once-daily
  * 100 kg and above: 7500 IU subcutaneously once-daily
  Other Names: dalteparin; Fragmin
  Arms: Low dose LMWH
Drug: Intermediate dose dalteparin — Intermediate weight-adjusted dose dalteparin:
  * < 50 kg: 7500 IU subcutaneously once-daily, or;
  * 50 kg to < 70 kg: 10000 IU subcutaneously once-daily, or;
  * 70 kg to < 100 kg: 12500 IU subcutaneously once-daily, or;
  * 100 kg or above: 15000 IU subcutaneously once-daily.
  Other Names: dalteparin; Fragmin
  Arms: Intermediate dose LMWH
Drug: Fixed low dose tinzaparin — Fixed low dose tinzaparin:
  * < 100 kg: 3500 IU subcutaneously once-daily
  * 100 kg and above: 4500 IU subcutaneously once-daily
  Other Names: tinzaparin; Innohep
  Arms: Low dose LMWH
Drug: Intermediate dose tinzaparin — Intermediate weight-adjusted dose tinzaparin:
  * < 50 kg: 4500 IU subcutaneously once-daily, or;
  * 50 kg to < 70 kg: 7000 IU subcutaneously once-daily, or;
  * 70 kg to < 100 kg: 10000 IU subcutaneously once-daily, or;
  * 100 kg or above: 12000 IU subcutaneously once-daily.
  Other Names: tinzaparin; Innohep
  Arms: Intermediate dose LMWH

SUMMARY:
This is a randomized-controlled open-label trial comparing two different doses of low-molecular-weight heparin (LMWH) in pregnant patients with a history of previous venous thromboembolism (VTE). Both doses are recommended doses in the 2012 guidelines of the American College of Chest Physicians (ACCP), but it is not known which dose is more efficacious in preventing recurrent venous thromboembolism in pregnancy.

Patients enter the study and will be randomized as soon as a home test confirms pregnancy. LMWH will be administered until 6 weeks postpartum. Follow-up will continue until 3 months postpartum. Patients will be recruited by their treating physician, either an obstetrician or internist.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years or older, and;
* Pregnancy confirmed by urinary pregnancy test, and;
* Gestational age < 14 weeks, and;
* Previous objectively confirmed VTE, either unprovoked, in the presence of use of oral contraceptives or estrogen/progestagen use, or related to pregnancy or the postpartum period, or minor risk factors (e.g. long distance travel, minor trauma).

Exclusion Criteria:

* Previous VTE related to a major provoking risk factor (e.g. surgery, major trauma or plaster cast immobilisation in the 3 months prior to VTE) as the sole risk factor, or;
* Indication for treatment with therapeutic dose anticoagulant therapy (e.g. treatment of acute VTE; permanent use of therapeutic anticoagulants outside of pregnancy), or;
* Inability to provide informed consent, or;
* Any contraindication listed in the local labelling of LMWH.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1110 (Actual)
Dates: Start 2013-04-24 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Symptomatic confirmed deep venous thrombosis | From date of randomization up to 6 weeks postpartum
  All events of symptomatic deep venous thrombosis in subjects will be recorded from the the date of randomization up to 6 weeks postpartum.
  Definition of symptomatic deep venous thrombosis (DVT):
  Suspected (recurrent) DVT with one of the following findings:
  If there were no previous DVT investigations:
  * Abnormal compression ultrasound (CUS),
  * An intraluminal filling defect on venography.
  If there was a previous DVT investigation:
  * Abnormal CUS where compression had been normal or, if non-compressible during screening, a substantial increase (4 mm or more) in diameter of the thrombus during full compression,
  * An extension of an intraluminal filling defect, or a new intraluminal filling defect or an extension of non-visualization of veins in the presence of a sudden cut-off on venography.
Symptomatic confirmed pulmonary embolism | From date of randomization up to 6 weeks postpartum
  All events of symptomatic pulmonary embolism in subjects will be recorded from the the date of randomization up to 6 weeks postpartum.
  Definition of symptomatic pulmonary embolism (PE):
  Suspected PE with one of the following findings:
  * A (new) intraluminal filling defect in subsegmental or more proximal branches on spiral CT scan
  * A (new) intraluminal filling defect or an extension of an existing defect or a new sudden cut-off of vessels more than 2.5 mm in diameter on the pulmonary angiogram
  * A (new) perfusion defect of at least 75% of a segment with a local normal ventilation result (high-probability) on ventilation/perfusion lung scan (VPLS)

SECONDARY OUTCOMES:
Symptomatic confirmed deep venous thrombosis | From date of randomization up to 3 months postpartum
  All events of symptomatic deep venous thrombosis in subjects will be recorded from the the date of randomization up to 3 months postpartum.
  Definition of symptomatic deep venous thrombosis (DVT):
  Suspected (recurrent) DVT with one of the following findings:
  If there were no previous DVT investigations:
  * Abnormal compression ultrasound (CUS),
  * An intraluminal filling defect on venography.
  If there was a previous DVT investigation:
  * Abnormal CUS where compression had been normal or, if non-compressible during screening, a substantial increase (4 mm or more) in diameter of the thrombus during full compression,
  * An extension of an intraluminal filling defect, or a new intraluminal filling defect or an extension of non-visualization of veins in the presence of a sudden cut-off on venography.
Symptomatic confirmed pulmonary embolism | From date of randomization up to 3 months postpartum
  All events of symptomatic pulmonary embolism in subjects will be recorded from the the date of randomization up to 3 months postpartum.
  Definition of symptomatic pulmonary embolism (PE):
  Suspected PE with one of the following findings:
  * A (new) intraluminal filling defect in subsegmental or more proximal branches on spiral CT scan
  * A (new) intraluminal filling defect or an extension of an existing defect or a new sudden cut-off of vessels more than 2.5 mm in diameter on the pulmonary angiogram
  * A (new) perfusion defect of at least 75% of a segment with a local normal ventilation result (high-probability) on ventilation/perfusion lung scan (VPLS)

OTHER OUTCOMES:
Major bleeding | During pregnancy until 3 months postpartum
  Major bleeding is defined as overt bleeding and:
  * Associated with a fall in hemoglobin of 2 g/dL or more, or
  * Leading to a transfusion of 2 or more units of packed red blood cells or whole blood, or
  * Occurring in a critical site: intracranial, intraspinal, intraocular, pericardial, intra-articular, intramuscular with compartment syndrome, retro-peritoneal, or
  * Contributing to death
Composite of major bleeding and clinically relevant non-major bleeding | During pregnancy until 3 months postpartum
  See 'Major bleeding' for the definition.
  Clinically relevant non-major bleeding is defined as overt bleeding not meeting the criteria for major bleeding but associated with medical intervention, unscheduled contact (visit or telephone call) with a physician, (temporary) cessation of study treatment, or associated with discomfort such as pain, or impairment of activities of daily life.
  * Hematuria if it is macroscopic, and either spontaneous or lasts for more than 24 hours after instrumentation (e.g. catheter placement or surgery) of the urogenital tract, or
  * Macroscopic gastro-intestinal haemorrhage: at least one episode of melena/hematemesis, if clinically apparent, or
  * Rectal blood loss, if more than a few spots, or
  * Hemoptysis, if more than a few speckles in the sputum, or
  * Intramuscular hematoma, or
  * Subcutaneous hematoma if the size is larger than 25 cm2, or larger than 100 cm2 if provoked, or
  * Multiple source bleeding
Early postpartum hemorrhage | Within 24 hours of delivery
  Postpartum haemorrhage is defined as blood loss of more than 500 mL within 24 hours of delivery (WHO-criteria). Severe postpartum haemorrhage is defined as blood loss of more than 1000 mL within 24 hours of delivery.
Blood transfusion < 6 weeks after delivery | Within 6 weeks of delivery
Blood transfusion < 24 hours postpartum | Within 24 hours of delivery
Late postpartum hemorrhage | From 24 hours postpartum to 6 weeks postpartum
  Postpartum haemorrhage is defined as blood loss of more than 500 mL within 24 hours of delivery (WHO-criteria). Severe postpartum haemorrhage is defined as blood loss of more than 1000 mL within 24 hours of delivery.
Mortality | During pregnancy until 3 months postpartum
Minor bleeding | During pregnancy until 3 months postpartum
  Minor bleeding is defined as all other overt bleeding episodes not meeting the criteria for major or clinically relevant bleeding or postpartum haemorrhage.
Skin complications | During pregnancy until 3 months postpartum
  e.g. itching, swelling, pain
Easy bruising | During pregnancy until 3 months postpartum
Necessity to switch to other LMWH | During pregnancy until 6 weeks postpartum
Heparin-induced thrombocytopenia | During pregnancy until 3 months postpartum
  Heparin-induced thrombocytopenia is defined according to the criteria of the ACCP guidelines.
Congenital anomalies or birth defects | During pregnancy until 3 months postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Saskia Middeldorp, MD PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (72):
- Weill Cornell Medicine | NewYork-Presbyterian, New York, New York, United States
- KU Leuven, Leuven, Belgium
- The Ottawa Hospital, Ottawa, Canada
- Denmark (2):
  - Aalborg University Hospital, Aalborg
  - Aarhus University Hospital, Aarhus
- France (23):
  - CHU de Besancon, Besançon
  - CHU de Bordeaux, Bordeaux
  - CHU de Brest, Brest
  - CHU de Caen, Caen
  - CHU de Clermont - Ferrand, Clermont-Ferrand
  - APHP Louis Mourier, Colombes
  - CHU de Grenoble, Grenoble
  - CHU de Limoges, Limoges
  - Hopiteaux de Marseille, Marseille
  - Marseille St Joseph, Marseille
  - CHU de Nancy, Nancy
  - CHU de Nice, Nice
  - CHU de Nîmes, Nîmes
  - APHP Antoine Béclère, Paris
  - APHP Port Royal, Paris
  - CHU de Poitiers, Paris
  - Centra Hospitalier de Roanne, Roanne
  - La Réunion - Saint-Denis, Saint-Denis
  - Hopital Nord, CHU de Saint Etienne, Saint-Etienne
  - La Réunion deSt Pierre, Saint-Pierre
  - Polyclinique de Sète, Sète
  - CHIC de Toulon, Toulon
  - CHU de Tours, Tours
- Ireland (6):
  - Corke University Hospital, Cork
  - Coombe Women's Hospital, Dublin
  - Rotunda Hospital, Dublin
  - The National Maternity Hospital, Dublin
  - Letterkenny University Hospital, Letterkenny
  - University Hospital Limerick, Limerick
- Netherlands (35):
  - Academic Medical Center, Amsterdam, North Holland
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Flevoziekenhuis, Almere Stad
  - OLVG oost, Amsterdam
  - SLAZ, Amsterdam
  - VU medical center, Amsterdam
  - Gelre Ziekenhuizen, Apeldoorn
  - Rijnstate hospital, Arnhem
  - Wilhelmina Ziekenhuis, Assen
  - Rode Kruis Ziekenhuis, Beverwijk
  - Amphia ziekenhuis, Breda
  - Reinier de Graaf Groep, Delft
  - Deventer Ziekenhuis, Deventer
  - Slingeland, Doetinchem
  - Albert Schweitzer, Dordrecht
  - Gelderse Vallei, Ede
  - Admiraal de Ruijter Ziekenhuis, Goes
  - Groene Hart Ziekenhuis, Gouda
  - Martini Ziekenhuis, Groningen
  - UMCG, Groningen
  - Spaarne Gasthuis, Haarlem
  - St Jansdal, Harderwijk
  - Atrium MC, Heerlen
  - MC Leeuwarden, Leeuwarden
  - LUMC, Leiden
  - MUMC, Maastricht
  - Canisius-Wilhelmina Ziekenhuis, Nijmegen
  - St. Radboud UMC, Nijmegen
  - Erasmus MC, Rotterdam
  - Bronovo ziekenhuis, The Hague
  - HAGA ziekenhuis, The Hague
  - TweeSteden, Tilburg
  - Diakonessen Utrecht, Utrecht
  - UMCU, Utrecht
  - Máxima MC, Veldhoven
- Oslo University Hospital, Oslo, Norway
- Federal State Institution "Research Center for Obstetrics, Gynecology and Perinatology", Moscow, Russia
- Vall d'Hebron Hospital, Barcelona, Spain

REFERENCES:
- [Background] Greer IA. Thrombosis in pregnancy: maternal and fetal issues. Lancet. 1999 Apr 10;353(9160):1258-65. doi: 10.1016/S0140-6736(98)10265-9. PMID 10217099
- [Background] Pabinger I, Grafenhofer H, Kyrle PA, Quehenberger P, Mannhalter C, Lechner K, Kaider A. Temporary increase in the risk for recurrence during pregnancy in women with a history of venous thromboembolism. Blood. 2002 Aug 1;100(3):1060-2. doi: 10.1182/blood-2002-01-0149. PMID 12130523
- [Background] White RH, Chan WS, Zhou H, Ginsberg JS. Recurrent venous thromboembolism after pregnancy-associated versus unprovoked thromboembolism. Thromb Haemost. 2008 Aug;100(2):246-52. PMID 18690344
- [Background] Bates SM, Greer IA, Middeldorp S, Veenstra DL, Prabulos AM, Vandvik PO. VTE, thrombophilia, antithrombotic therapy, and pregnancy: Antithrombotic Therapy and Prevention of Thrombosis, 9th ed: American College of Chest Physicians Evidence-Based Clinical Practice Guidelines. Chest. 2012 Feb;141(2 Suppl):e691S-e736S. doi: 10.1378/chest.11-2300. PMID 22315276
- [Background] Greer IA, Nelson-Piercy C. Low-molecular-weight heparins for thromboprophylaxis and treatment of venous thromboembolism in pregnancy: a systematic review of safety and efficacy. Blood. 2005 Jul 15;106(2):401-7. doi: 10.1182/blood-2005-02-0626. Epub 2005 Apr 5. PMID 15811953
- [Background] Tooher R, Gates S, Dowswell T, Davis LJ. Prophylaxis for venous thromboembolic disease in pregnancy and the early postnatal period. Cochrane Database Syst Rev. 2010 May 12;(5):CD001689. doi: 10.1002/14651858.CD001689.pub2. PMID 20464719
- [Background] Sanson BJ, Lensing AW, Prins MH, Ginsberg JS, Barkagan ZS, Lavenne-Pardonge E, Brenner B, Dulitzky M, Nielsen JD, Boda Z, Turi S, Mac Gillavry MR, Hamulyak K, Theunissen IM, Hunt BJ, Buller HR. Safety of low-molecular-weight heparin in pregnancy: a systematic review. Thromb Haemost. 1999 May;81(5):668-72. PMID 10365733
- [Background] Lepercq J, Conard J, Borel-Derlon A, Darmon JY, Boudignat O, Francoual C, Priollet P, Cohen C, Yvelin N, Schved JF, Tournaire M, Borg JY. Venous thromboembolism during pregnancy: a retrospective study of enoxaparin safety in 624 pregnancies. BJOG. 2001 Nov;108(11):1134-40. doi: 10.1111/j.1471-0528.2003.00272.x. PMID 11762651
- [Background] Pabinger I, Grafenhofer H, Kaider A, Kyrle PA, Quehenberger P, Mannhalter C, Lechner K. Risk of pregnancy-associated recurrent venous thromboembolism in women with a history of venous thrombosis. J Thromb Haemost. 2005 May;3(5):949-54. doi: 10.1111/j.1538-7836.2005.01307.x. PMID 15869590
- [Background] Roeters van Lennep JE, Meijer E, Klumper FJ, Middeldorp JM, Bloemenkamp KW, Middeldorp S. Prophylaxis with low-dose low-molecular-weight heparin during pregnancy and postpartum: is it effective? J Thromb Haemost. 2011 Mar;9(3):473-80. doi: 10.1111/j.1538-7836.2011.04186.x. PMID 21232006
- [Background] Lindqvist PG, Bremme K, Hellgren M; Working Group on Hemostatic Disorders (Hem-ARG), Swedish Society of Obstetrics and Gynecology. Efficacy of obstetric thromboprophylaxis and long-term risk of recurrence of venous thromboembolism. Acta Obstet Gynecol Scand. 2011 Jun;90(6):648-53. doi: 10.1111/j.1600-0412.2011.01098.x. Epub 2011 Apr 15. PMID 21314819
- [Background] Roshani S, Cohn DM, Stehouwer AC, Wolf H, van der Post JA, Buller HR, Kamphuisen PW, Middeldorp S. Incidence of postpartum haemorrhage in women receiving therapeutic doses of low-molecular-weight heparin: results of a retrospective cohort study. BMJ Open. 2011 Nov 14;1(2):e000257. doi: 10.1136/bmjopen-2011-000257. Print 2011. PMID 22102641
- [Background] Kaandorp SP, Goddijn M, van der Post JA, Hutten BA, Verhoeve HR, Hamulyak K, Mol BW, Folkeringa N, Nahuis M, Papatsonis DN, Buller HR, van der Veen F, Middeldorp S. Aspirin plus heparin or aspirin alone in women with recurrent miscarriage. N Engl J Med. 2010 Apr 29;362(17):1586-96. doi: 10.1056/NEJMoa1000641. Epub 2010 Mar 24. PMID 20335572
- [Derived] Bistervels IM, Wiegers HMG, Ainle FN, Bleker SM, Chauleur C, Donnelly J, Jacobsen AF, Rodger MA, DeSancho MT, Verhamme P, Hansen AT, Shmakov RG, Ganzevoort W, Buchmuller A, Middeldorp S; Highlow Investigators. Onset of labor and use of analgesia in women using thromboprophylaxis with 2 doses of low-molecular-weight heparin: insights from the Highlow study. J Thromb Haemost. 2023 Jan;21(1):57-67. doi: 10.1016/j.jtha.2022.11.004. Epub 2022 Dec 22. PMID 36695396
- [Derived] Bistervels IM, Buchmuller A, Wiegers HMG, Ni Ainle F, Tardy B, Donnelly J, Verhamme P, Jacobsen AF, Hansen AT, Rodger MA, DeSancho MT, Shmakov RG, van Es N, Prins MH, Chauleur C, Middeldorp S; Highlow Block writing committee; Highlow Investigators. Intermediate-dose versus low-dose low-molecular-weight heparin in pregnant and post-partum women with a history of venous thromboembolism (Highlow study): an open-label, multicentre, randomised, controlled trial. Lancet. 2022 Nov 19;400(10365):1777-1787. doi: 10.1016/S0140-6736(22)02128-6. Epub 2022 Oct 28. PMID 36354038
- [Derived] Middleton P, Shepherd E, Gomersall JC. Venous thromboembolism prophylaxis for women at risk during pregnancy and the early postnatal period. Cochrane Database Syst Rev. 2021 Mar 29;3(3):CD001689. doi: 10.1002/14651858.CD001689.pub4. PMID 33779986
- [Derived] Middeldorp S. New studies of low-molecular-weight heparin in pregnancy. Thromb Res. 2015 Feb;135 Suppl 1:S26-9. doi: 10.1016/S0049-3848(15)50436-2. Epub 2015 Feb 9. PMID 25903529
- [Derived] Bleker SM, Coppens M, Middeldorp S. Sex, thrombosis and inherited thrombophilia. Blood Rev. 2014 May;28(3):123-33. doi: 10.1016/j.blre.2014.03.005. Epub 2014 Apr 1. PMID 24768093